CLINICAL TRIAL: NCT01554579
Title: A Four-Week Multicenter Study Evaluating the Safety and Efficacy of Gefapixant (AF-219/MK-7264) in Subjects With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7264-004; AF219004 (Other: Afferent Pharmaceuticals)
Record Dates: First submitted 2012-03-12; First posted 2012-03-15 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Gefapixant; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar Pill
- Gefapixant (Experimental)
  Interventions: Drug: Gefapixant

INTERVENTIONS:
Drug: Gefapixant — BID
  Other Names: AF-219; MK-7264
  Arms: Gefapixant
Drug: Sugar Pill — Placebo
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to assess the efficacy of a single dose level of gefapixant (AF-219/MK-7264) in subjects with moderate to severe pain associated with osteoarthritis (OA) of the knee compared with placebo after 4 weeks of treatment.

The study will also assess the safety and tolerability, changes in physical function, stiffness, treatment response and health outcomes.

DETAILED DESCRIPTION:
Subjects who satisfy entry criteria at Screening will enter the Washout Phase, discontinuing their current nonsteroidal anti-inflammatory drug (NSAID) therapy.

Up to 220 subjects who fulfill flare (and other entry) criteria will be randomized to gefapixant or placebo.

Subjects will complete Treatment Visits 1, 2, 3, and 4 weeks after starting study drug. At each Treatment Visit, subjects will undergo efficacy assessments and safety procedures. During the Washout and Treatment Phases subjects will complete the 'average pain' Numeric Pain Rating Scale (NPRS) and count of rescue medication used for the preceding 24 hours.

Subjects will return 2 weeks after their last Treatment Visit (for a Follow-Up Visit).

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Women of child bearing potential must not be pregnant during the study and must use two forms of birth control
* Men and their female partners must use two forms of birth control
* Clinical and radiographic evidence of chronic knee osteoarthritis
* An average NPRS score of >=5 and <=9 over a 4-7 day washout period of their previous osteoarthritis medications
* Ambulatory
* Have provided written informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2012-03-29 (Actual); Primary Completion 2013-11-11 (Actual); Study Completion 2013-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Afferent Investigative Site, Phoenix, Arizona
  - Afferent Investigative Site, San Diego, California
  - Afferent Investigative Site, Clearwater, Florida
  - Afferent Investigative Site, Orlando, Florida
  - Afferent Investigative Site, Pinellas Park, Florida
  - Afferent Investigative Site, Atlanta, Georgia
  - Afferent Investigative Site, Wichita, Kansas
  - Afferent Investigative Site, New Bedford, Massachusetts
  - Afferent Investigative Site, Watertown, Massachusetts
  - Afferent Investigative Site, Troy, Michigan
  - Afferent Investigative Site, Olive Branch, Mississippi
  - Afferent Investigative Site, Hazelwood, Missouri
  - Afferent Investigative Site, St Louis, Missouri
  - Afferent Investigative Site, Albuquerque, New Mexico
  - Afferent Investigative Site, Asheville, North Carolina
  - Afferent Investigative Site, Greensboro, North Carolina
  - Afferent Investigative Site, Winston-Salem, North Carolina
  - Afferent Investigative Site, Cincinnati, Ohio
  - Afferent Investigative Site, Toledo, Ohio
  - Afferent Investigative Site, Medford, Oregon
  - Afferent Investigative Site, Duncansville, Pennsylvania
  - Afferent Investigative Site, Warwick, Rhode Island
  - Afferent Investigative Site, Greer, South Carolina
  - Afferent Investigative Site, Mt. Pleasant, South Carolina
  - Afferent Investigative Site, Austin, Texas
  - Afferent Investigative Site, Dallas, Texas
  - Afferent Investigative Site, Houston, Texas
  - Afferent Investigative Site, San Antonio, Texas
  - Afferent Investigative Site, Clinton, Utah
  - Afferent Investigative Site, Roanoke, Virginia
  - Afferent Investigative Site, Renton, Washington
  - Afferent Investigative Site, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Pill: Sugar Pill: Placebo Subjects in the trial received one tablet twice daily for 4 weeks.
- Gefapixant: Gefapixant: BID Subjects received one tablet twice daily for 4 weeks.
Period: Overall Study
Arm/Group | Sugar Pill | Gefapixant
Started | 86 | 85
Completed | 76 | 58
Not Completed | 10 | 27
Not completed — Adverse Event | 6 | 25
Not completed — Lack of Efficacy | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Gefapixant | Total
Number analyzed (Participants) | 86 | 85 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 65 | 129
  >=65 years | 22 | 20 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 57 | 109
  Male | 34 | 28 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 20 | 41
  White | 62 | 62 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 86 | 85 | 171
Numeric Pain Rating Scale (NPRS) [Mean (Full Range); unit: units on a scale] — Subjects were instructed to select a number between 0 and 10 where 0 is no pain and 10 is the worst possible pain. The scale was completed by telephone (an interactive voice response system [IVRS]) every evening before bedtime.
  units on a scale | 6.7 [5 to 9] | 6.8 [5 to 9] | 6.75 [5 to 9]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint of This Study is the Weekly Average Daily NPRS (Average Pain)
Description: Subjects were instructed to select a number on a scale that best described their knee arthritis pain during the past 24 hours. The scale was between 0 and 10 where 0 was no pain and 10 was the worst possible pain. The scale was completed by telephone (an interactive voice response system [IVRS]) every evening before bedtime.
Time Frame: 2 Weeks
Population: Per protocol population defined as subjects who received at least 1 dose of drug, had at least 1 post-baseline efficacy measure, complied with protocol and did not have major protocol deviations. Compliance with the protocol defined as having (in the last week of the study) a weekly average NPRS score w/ at least 50% non-missing dairy NPRS scores.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Sugar Pill | Gefapixant
Number analyzed (Participants) | 82 | 74
units on a scale | 5.3 [0 to 10] | 4.9 [0 to 10]

2. Secondary Outcome: WOMAC Scores
Description: This is the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). This is a questionnaire that asks subjects to evaluate their pain, stiffness, and physical activities affecting their knee over the past 48 hours. Subjects evaluate their pain, stiffness and physical activities by selecting a number between 0 and 10 where 0 is no pain/no stiffness/no difficulty doing physical activities and 10 is extreme pain/extreme stiffness/extreme difficulty doing physical activities. The questionnaire was administered at Screening, Baseline and at the end of Week 4 by telephone (an interactive voice response system [IVRS]) before bedtime. The scores for each category are totaled (range is 0-100). A lower total score means less pain and a higher total score means greater pain.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Gefapixant
Number analyzed (Participants) | 79 | 71
units on a scale | 40.7 (23.12) | 41.0 (25.26)

3. Secondary Outcome: SF-36
Description: The SF-36 (acute version 2) was a 36 question survey administered at Baseline and at the end of study or early termination (Week 4). The questionnaire contained numerous domain scores to evaluate physical function, mental function, general health, bodily pain, social functioning and vitality. The question of interest for the analysis was question #1 regarding walking pain. Scores range from 0 - 100. A lower score means decreased pain while walking and a higher score means increased pain while walking.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Gefapixant
Number analyzed (Participants) | 80 | 73
units on a scale | 3.8 (2.39) | 4.1 (2.77)

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Gefapixant
Serious Adverse Events (participants affected / at risk) | 1/86 | 0/85
Other Adverse Events (participants affected / at risk) | 17/86 | 75/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=86) | Gefapixant (N=85)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=86) | Gefapixant (N=85)
Dysgeusia (Nervous system disorders) | 4 (4) | 64 (64)
Ageusia (Nervous system disorders) | 0 (0) | 12 (12)
headache (Nervous system disorders) | 10 (10) | 9 (9)
hypogeusia (Nervous system disorders) | 0 (0) | 7 (7)
dizziness (Nervous system disorders) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
60 days prior to the submission of any results, the PI shall submit to SPONSOR any proposed PUBLICATION, which period may be extended for an additional 30 days if requested by SPONSOR. If any Confidential Information should be redacted or patent applications relating to an Invention should be filed prior to PUBLICATION, then PUBLICATION will be delayed until patent application has been filed. Delay of a PUBLICATION shall not exceed 24 months from the date of such notice to the PI.